CLINICAL TRIAL: NCT04038775
Title: Take 2 Pills and Go Volunteer in the Morning: A Feasibility Study of Engaging Patients as Volunteers
Brief Title: Take 2 Pills and Go Volunteer in the Morning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Julie Darnell, Associate Professor, Loyola University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 210989
Record Dates: First submitted 2019-05-29; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Volunteers
Keywords: medically uninsured

STUDY DESIGN:
Intervention Model Description: The first 25 patients are placed into the intervention group (recommended volunteering by their provider) and the next 25 patients are placed into the control group (not recommended volunteering).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volunteering (Experimental): The experimental arm will receive a volunteer "prescription" from their provider and assistance from a study team member to find a volunteer job.
  Interventions: Behavioral: Volunteering
- Control (No Intervention): The control arm will not be recommended to volunteer or assisted in finding a volunteer activity. They will answer the same survey questions as the intervention subjects.

INTERVENTIONS:
Behavioral: Volunteering — Subjects recommended volunteer by their provider.
  Arms: Volunteering

SUMMARY:
In this study, doctors will "prescribe" volunteer work for their patients. The investigators are determining whether it is feasible for providers to recommend volunteering to their patients, and whether patients who are recommended this "treatment" actually do volunteer work (i.e., find it "acceptable"). The study is focused on uninsured patients at Loyola Medicine's Access to Care (ATC) Clinic. The study's secondary aim is to determine whether or not engaging in volunteer work yields health benefits.

DETAILED DESCRIPTION:
In this feasibility study, doctors will "prescribe" volunteer work for their patients. The setting is Loyola Medicine's Access to Care Clinic, which serves patients who are low-income and uninsured (and often members of racial/ethnic minority groups). The investigators are determining whether it is feasible for providers in a low-resourced primary care setting to recommend volunteering to their patients, and whether patients who are recommended this "treatment" actually do volunteer work (and how much). The investigators are also interested in measuring whether volunteering is associated with any potential health benefits, specifically well-being and self-esteem.

Promoting volunteerism is the intervention because research evidence suggests that volunteer work may be good for one's health. For example, research shows that volunteering is associated with numerous potential health benefits: improved mental health, increased physical activity, higher preventive health care utilization, lower cardiovascular risk and lower mortality. Besides better health, volunteering also can teach valuable skills, help individuals meet others, and foster new relationships.

Despite all these potential benefits, rates of volunteering are low. Overall, just one in four people volunteers. Additionally, people who have lower incomes are less likely to volunteer (14% of people with incomes below $20,000 vs. 35% of people with incomes above $100,000. And minority groups are less likely to volunteer than whites (just 19% of African Americans and 15% of Latinos compared with 26% of Whites).

Thus, the intervention is aimed to increase volunteer participation rates among groups unlikely to volunteer: low-income uninsured persons who are members of racial/ethnic minority groups.

ELIGIBILITY:
Inclusion Criteria * Access to Care patient

Exclusion Criteria

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Total volunteer hours | Baseline to six months
  Investigators will sum the reported volunteer hours, which will be tracked at baseline and monthly for 6 months.

SECONDARY OUTCOMES:
Change in Rosenberg Self-Esteem Scale Score | Baseline to six months
  Using the Rosenberg Self-Esteem Scale, investigators will compare changes in the total score from baseline to six months. The minimum score is 10 and the maximum score is 40. Higher scores indicate a better outcome, i.e, higher self-esteem. The Rosenberg Self-Esteem Scale is administered twice: at baseline and at six months after baseline.
Change in Patient-Reported Outcome Measurement Information System (PROMIS) Global Health Short Form Scale | Baseline to six months
  Using the PROMIS Global Health Short Form Scale, investigators will compare changes in the physical and mental subscores from baseline to six months. Higher scores reflect a better outcome, i.e., better functioning. The range of both the physical and mental health subscales range from 2 to 10. Raw scores will be converted to t-scores to facilitate interpretation. The PROMIS Global Health Short Form is administered twice: at baseline and at six months after baseline.
Change in the Arizona Integrative Outcomes Scale | Baseline to six months
  Using the Arizona Integrative Outcomes Scale (AIOS), a visual analogue measure of well-being, investigators will compare changes from baseline to six months. Scores range from 0 to 100, with higher scores reflecting a better outcome, i.e., better well-being.The AIOS is administered twice: at baseline and at six months after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Julie S Darnell, PhD, Principal Investigator — Loyola University Chicago
Locations (1):
- Access to Care Clinic, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
This is a feasibility study. There are no plans to share data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT04038775/Prot_SAP_000.pdf